CLINICAL TRIAL: NCT02587208
Title: Plastibell Versus Conventional Dissection Techniques for Circumcision in Infants
Brief Title: Plastibell Versus Conventional Dissection Techniques for Circumcision in Infants and Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr Abdulrahman Alzahem, Associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E14-1270
Record Dates: First submitted 2015-08-30; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Circumcision, Male
Keywords: circumcision; plastibell; infants; open sleeve

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional sleeve (Active Comparator): In the sleeve dissection group, a double incision technique on both outer and inner layers of the foreskin is employed. Hemostasis is achieved by bipolar diathermy, and cut edges are sutured with 5/0 rapide vicryl.
  Interventions: Procedure: conventional sleeve
- plastibell (Active Comparator): In the Plastibell group, the size of the device is chosen according to the lateral-lateral diameter of the glans. A dorsal slit incision is made and then the foreskin is pulled up and the Plastibell device placed between the prepuce and the glans. A non-absorbable string was tightly tied around the device and the distal prepuce is removed.
  Interventions: Device: Plastibell

INTERVENTIONS:
Device: Plastibell — In the Plastibell group, the size of the device is chosen according to the lateral-lateral diameter of the glans. A dorsal slit incision is made and then the foreskin is pulled up and the Plastibell device placed between the prepuce and the glans. A non-absorbable string was tightly tied around the device and the distal prepuce is removed.
  Arms: plastibell
Procedure: conventional sleeve — In the sleeve dissection group, a double incision technique on both outer and inner layers of the foreskin is employed. Hemostasis is achieved by bipolar diathermy, and cut edges are sutured with 5/0 rapide vicryl.
  Arms: conventional sleeve

SUMMARY:
Outcome of circumcision with Plastibell or conventional dissection techniques in infants and children: A prospective randomized controlled trial

Aim: to evaluate and compare postoperative and esthetic outcomes after Plastibell and conventional dissection circumcision

Methods:

Randomized Controlled Trial Inclusion criteria: patients younger than 13 years including neonates who required circumcision for various indications.

Exclusion criteria: - patients with bleeding or clotting disorders

* Those whose parents insisted on a particular type of surgery
* Children with lateral- lateral diameter of the glans over which a Plastibell device could not be placed Primary endpoint: parental concerns and satisfaction (questionnaire) Secondary endpoints: composite morbidity, operative time, postoperative pain (analgesic requirements)
* Early postoperative problems: infection, bleeding, swelling, dysuria, pain (incidence, mean duration, emergency care if necessary, parental concerns about them (on a Likert-type 5-point scale [ not at all, a little, rather, very, very much])
* Irregular scar, jumbling of tissues at the site of frenulum (assessed by physician)
* Postoperative adhesions (assessed by physician)
* Postoperative pain and analgesic requirements (paracetamol 15 mg/kg PO Q6 hrs for 48 hrs then PRN) number of doses and days required for analgesia as judged by parents, VAS ( >- 6 SCORE ), Kaplan-Meier analysis (time to event)
* Parental satisfaction ( overall esthetic outcome [ very much satisfied, very satisfied, rather, a little satisfied, not at all satisfied])
* Parental satisfaction ( skin removal): excess skin removal, insufficient skin removal [ not at all, a little, rather, very, very much]
* Time for bell separation (mean +-SD), Kaplan-Meier analysis for different age groups

DETAILED DESCRIPTION:
Outcome of circumcision with Plastibell or conventional dissection techniques in infants and children: A prospective randomized controlled trial Aim: to evaluate and compare postoperative and esthetic outcomes after Plastibell and conventional dissection circumcision

Methods:

A balanced, parallel group, prospective randomized controlled trial is to be performed over 2 years at our institute. Patients enrollment will commence after approval of our institutional review board as well as obtaining informed consent from the patient's legal guardians.

Participants Inclusion criteria: Patients younger than 13 years including neonates who required circumcision for various indications.

Exclusion criteria: - Patients with bleeding or clotting disorders

* Patients with hypospadias or other penile anomalies
* Those whose parents insisted on a particular type of surgery
* Children with lateral- lateral diameter of the glans over which a Plastibell device could not be placed Interventions The subjects will be randomized and allocated into two groups: the Plastibell and sleeve dissection techniques.

Sample size calculation Power calculation was based on aesthetic outcome which was based on previous studies (Nagdeve et al and Fraser et al) wherein 60-69% of subjects operated by Plastibell technique and 43-45% by conventional dissection technique had good satisfaction. Establishing alpha at 0.2 and a power of 0.80 produced a sample size of 50 patients per arm.

Assignment and randomization A block randomization scheme will be used with equal allocation of subjects to the Plastibell and sleeve dissection groups. There are a total of 10 blocks, each having 10 subjects. One block will be selected by simple random sampling and its subjects will be subjected to the intervention.

Protocol All the parents will be informed regarding details of surgery, complications, postoperative care and follow-up protocol. Both procedures are performed under light general anesthesia and either dorsal penile nerve block or caudal block. The first step in both groups is to separate the foreskin from the glans penis and removal of smegma.

In the Plastibell group, the size of the device is chosen according to the lateral-lateral diameter of the glans. A dorsal slit incision is made and then the foreskin is pulled up and the Plastibell device placed between the prepuce and the glans. A non-absorbable string was tightly tied around the device and the distal prepuce is removed.

In the sleeve dissection group, a double incision technique on both outer and inner layers of the foreskin is employed. Hemostasis is achieved by bipolar diathermy, and cut edges are sutured with 5/0 rapide vicryl.

All patients will be managed on a day-care basis. At discharge, they will be prescribed syrup/tablet paracetamol 15mg/kg/dose every 6 hours whenever needed if pain score >_6 based on a visual analog scale for pain assessment. Parents will be told to write down how many times they give analgesic each day until the first postoperative visit.

Follow-up will be done at 14th (or after separation of Plastibell whichever later) and 90th days after surgery.

Written questionnaires will be given to parents at time of discharge Primary endpoint: Parental concerns and satisfaction (questionnaire) Secondary endpoints: Composite Morbidity, Operative Time, Postoperative Pain (analgesic requirements)

* Early postoperative problems: infection, bleeding, swelling, dysuria, pain (incidence, mean duration, emergency care if necessary, parental concerns about them (on a Likert-type 5-point scale [not at all, a little, rather, very, very much])
* Irregular scar, jumbling of tissues at the site of frenulum (assessed by physician)
* Postoperative adhesions (assessed by physician)
* Postoperative pain and analgesic requirements (paracetamol 15 mg/kg PO Q6 hrs PRN) number of doses and days required for analgesia as judged by parents, VAS ( >- 6 SCORE ), Kaplan-Meier analysis (time to event)
* Parental satisfaction ( overall esthetic outcome [ very much satisfied, very satisfied, rather, a little satisfied, not at all satisfied])
* Parental satisfaction ( skin removal): excess skin removal, insufficient skin removal [ not at all, a little, rather, very, very much]
* Time for bell separation (mean +-SD), Kaplan-Meier analysis for different age groups

ELIGIBILITY:
Inclusion Criteria:

* Patients 3 months - 12 years (inclusive) who required circumcision for various indications.

Exclusion Criteria:

* Patients with bleeding or clotting disorders
* Those whose parents insisted on a particular type of surgery
* Children with lateral- lateral diameter of the glans over which a Plastibell device could not be placed

Ages: 3 Months to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Questionnaire for Parental satisfaction (overal esthetic outcome) | 3-6 months
  - Parental satisfaction ( overall esthetic outcome [ very much satisfied, very satisfied, rather, a little satisfied, not at all satisfied])

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Postoperative pain measures | 1-2 weeks
  VAS ( >6/10) score would entitle giving paracetamol for patient and the total doses/total days where paracetamol was needed will be calculated
Early composite morbidity (incidence % and mean duration) | 2-4 weeks
  Early postoperative problems: infection, bleeding, swelling, dysuria, pain (incidence, mean duration, emergency care if necessary
Likert -type 5-point scale for Parental concerns about early composite morbidity | 2-4 weeks
  parental concerns about them (on a Likert-type 5-point scale [not at all, a little, rather, very, very much])

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Alzahem, MBBS, FRCSC, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Riyadh Region, Saudi Arabia